CLINICAL TRIAL: NCT00279032
Title: A Randomised, Placebo-Controlled, Double-Blind, Parallel Group Study to Investigate the Effects of Chronic Dose Oral GW406381 on Pain and Areas of Hyperalgesia and Allodynia in Patients With Peripheral Nerve Injury as a Result of Trauma or Surgery.
Brief Title: GW406381 In Patients With Peripheral Nerve Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CXA10006
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2009-02-23 (Estimated); Status verified 2009-02

CONDITIONS: Hyperalgesia; Neurodynia; Pain; Trauma
Keywords: GW406381; peripheral nerve injury; patients; allodynia; hyperalgesia; randomised; placebo-controlled
MeSH Terms: conditions — Hyperalgesia; Neuralgia; Pain; Wounds and Injuries; Peripheral Nerve Injuries | interventions — GW406381X

INTERVENTIONS:
Drug: GW406381

SUMMARY:
The findings from preclinical animal models confirm the peripheral anti-inflammatory/analgesic activity of GW406381 and also suggest contribution of a central site of action to the anti-hyperalgesic efficacy that may not be shared by other COX-2 inhibitors. A central action is consistent with distribution of GW406381 into the CNS in animals. Furthermore, preliminary data from a positron emission tomography study in which 6 healthy male volunteers received a tracer dose of 11C labelled GW406381 indicate that GW406381 is rapidly absorbed into the central nervous system in man.

ELIGIBILITY:
Inclusion criteria:

* Baseline average daily Pain Score of greater than or equal to 4 (averaged over the 7 days prior to Treatment Visit 1), as reported on the 11 point pain intensity numerical rating scale.
* Subjects on medications for neuropathic pain or received nerve blocks for neuropathic pain.

Exclusion criteria:

* Known history of hypersensitivity or intolerance to acetaminophen, paracetamol, aspirin, COX-2 inhibitors or NSAIDs.
* Subject is unable to discontinue NSAIDs or COX-2 inhibitors (except aspirin as a cardioprotective; certain doses apply), topical lidocaine and topical capsaicin for the treatment of pain for the period prior to randomization and for the duration of the study.
* Subject is unable to refrain from sedative use during the study (benzodiazepines prescribed as hypnotic sleep agents allowed).
* Subject is unable to refrain from nerve blocks for 4 weeks prior to randomisation and during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-09

PRIMARY OUTCOMES:
To investigate the effect of chronic oral dosing (21 days) of GW406381 compared to placebo, on pain in patients with peripheral nerve injury

SECONDARY OUTCOMES:
To investigate the effect of 21 days oral dosing of GW406381 on thermal hyperalgesia, dynamic allodynia and static mechanical hyperalgesia in patients with peripheral nerve injury.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (5):
- United Kingdom (5):
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Liverpool, Lancashire
  - GSK Investigational Site, Leicester, Leicestershire
  - GSK Investigational Site, Solihull, West Midlands
  - GSK Investigational Site, London